CLINICAL TRIAL: NCT07275138
Title: Acute Cardiovascular and Neuromuscular Responses to Walking With Blood Flow Restriction in Older Adults: a Study Protocol for a Randomized Crossover Trial
Brief Title: Acute Cardiovascular and Neuromuscular Responses to Walking With Blood Flow Restriction (BFR) in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Ministry of Work and Welfare - Xunta de Galicia (Other Government); Universidade do Porto (Other); University of La Laguna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CEFADE40_2024; ED481B-2024/079 (Other Grant/Funding Number: Xunta de Galicia)
Record Dates: First submitted 2025-11-17; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy Older Adults
Keywords: Blood Flow Restriction (BFR); walking exercise; older adults; Gait Kinematic; Cardiovascular Response; Neuromuscular Performance; Crossover Study; Physical Function; safety; Endurance training; Low-impact exercise; Aerobic exercise; Physical activity; functionality; Elderly; Senior; Age 60+; Community-dwelling; Non-institutionalized; Partial Blood Flow Restriction; Limb Occlusion Training; Vascular Occlusion Training; KAATSU Training; Low-load resistance training with BFR; Occlusion exercise; walking; walking training; exercise training
MeSH Terms: conditions — Motor Activity | interventions — Walking; Exercise

STUDY DESIGN:
Intervention Model Description: Each participant will perform a walking experimental session under different levels of BFR applied to the lower limbs. The order of BFR conditions will be randomized for each participant. A minimum washout period of 72 hours will be observed between sessions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of the condition for each session. One researcher sets the BFR, while a second, blinded researcher supervises and assesses the participant. Data will be analyzed by an external analyst using coded data, keeping session conditions unknown.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BFR40% (Experimental): BFR set at 40% of the participant's arterial occlusion pressure (AOP).
  Interventions: Behavioral: Walking
- BFR80% (Experimental): BFR set at 80% of the participant's AOP.
  Interventions: Behavioral: Walking
- BFR0% (Sham Comparator): BFR set at 0% of the participant's AOP.
  Interventions: Behavioral: Walking
- CON (Active Comparator): No BFR cuffs.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Participants will perform two continuous 10-minute walking bouts, separated by a 3-minute seated recovery period to allow reperfusion following BFR or pause, along a rectangular 40-meter walking circuit (15×5 m). Walking cadence will be standardized at 112 steps per minute.
  Other Names: Physical activity; Aerobic exercise; Cardio exercise; Endurance exercise; Functional movement

SUMMARY:
The goal of this clinical trial is to explore how walking combined with different levels of partial blood flow restriction (BFR) affects cardiovascular, neuromuscular, and movement (kinematic) variables in older adults.

The main questions it aims to answer are:

Does walking with BFR increase internal effort, as shown by cardiovascular changes, and is this effect proportional to the level of restriction?

Does walking with BFR temporarily reduce neuromuscular control, and is this reduction greater at higher restriction levels?

Does walking with BFR change gait movement patterns?

This study uses a crossover design, meaning that each participant will complete all four conditions and serve as their own control.

Participants will:

Take part in walking sessions under four conditions with different levels of restriction: BFR40%, BFR80%, SHAM (0% BFR), and CON (without BFR).

Have their cardiovascular responses, muscle performance, and gait movement patterns measured.

Report their perceptions of the sessions, including Rate of Perceived Exertion (RPE), satisfaction, and possible side effects.

DETAILED DESCRIPTION:
This innovative research project aims to explore the effect of the novel BFR technique, combined with walking, as a non-pharmacological strategy to prevent or reverse sarcopenia and thereby improve the quality of life in sedentary older adults. BFR involves the use of a specialized pneumatic cuff to restrict venous blood flow to a muscle while partially inhibiting arterial flow, and it can be applied either at rest or in combination with exercise.

The application of BFR combined with exercise has shown promise as a tool to induce favorable physiological effects at lower training doses, that is, at lower intensities (e.g., lower intensities or slower walking or running speeds), compared to active control groups. However, despite the promising benefits reported in some studies, comprehensive investigation of the cardiovascular and neuromuscular responses during BFR combined with walking remains a largely unexplored area, both in healthy participants and special populations. This knowledge gap is particularly relevant when considering the substantial benefits that older adults and individuals with mobility limitations could gain from BFR combined with walking, especially given their potential difficulty in adhering to the minimum exercise dosage requirements recommended by the World Health Organization

ELIGIBILITY:
Inclusion Criteria:

• Aged between 60 and 90 years.

Exclusion Criteria:

* Being institutionalized.
* Peripheral vascular disease, defined by an ankle-brachial index (ABI) outside the normal range (0.9-1.4).
* Uncontrolled arterial hypertension (>180/110 mmHg).
* Any contraindication to exercise, based on self-reported medical history and PAR-Q+.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 25 minutes
  Systolic, diastolic and mean blood pressure will be obtained by a photoplethysmography sensor. Units: mmHg
Heart rate | 60 minutes
  The average and maximum values will be obtained using a chest-worn heart rate sensor. Unit: beats per minute (bpm)
RR-Interval Time-Domain Metrics | 60 minutes
  Standard time-domain HRV metrics-including mean RR intervals (meanRR), the standard deviation of normal-to-normal intervals (SDNN), and the root mean square of successive differences (RMSSD)-will be derived from inter-beat interval data exported from a chest-worn heart rate sensor (epochs of 5 min).
  Units: milliseconds (ms).
RR-Interval Nonlinear Metric | 60 minutes
  Short-term fractal scaling (DFA α1) will be calculated from inter-beat interval data exported from a chest-worn heart rate sensor (epochs of 5 min).
  Units: dimensionless.
Maximum isometric strength | 10 minutes
  Maximum voluntary isometric contraction (MVIC) force during a knee-extension task will be recorded using a force-gauge device.
  Unit: Newtons (N)
Force steadiness | 10 minutes
  Force steadiness will be evaluated from the RMSSD of the coefficient of variation (CV) during a 30-s submaximal isometric knee-extension contraction at 30% MVIC, using a force-gauge device with data-analysis software.
  Unit: Percentage (%)

SECONDARY OUTCOMES:
Arterial stiffness | 25 minutes
  It will be assessed by finger-toe pulse wave velocity (PWV) method. Units: m/s
Temporal Gait Parameters | 20 minutes
  Mean temporal gait parameters-including stride time, step time, and stance time-will be derived from IMU-based measurements.
  Units: milliseconds (ms).
Temporal Gait Variability | 20 minutes
  Stride-to-stride temporal variability (stride time, step time, stance time) will be computed from walking recordings collected using a wearable inertial measurement unit (IMU) equipped with a triaxial accelerometer and gyroscope. Variability will be expressed as the coefficient of variation (CV) for each temporal metric.
  Units: Percentage (%)
Postural Stability | 10 minutes
  Postural stability in mediolateral (ML) and anterior-posterior (AP) directions will be assessed during quiet standing under four conditions (eyes open/closed × firm/foam surface). A wearable IMU will record triaxial centre-of-mass acceleration. Stability metrics will be computed as -ln[m/s²], where higher values reflect lower acceleration and therefore better postural control.
  Units: -ln[m/s²]
Internal subjective load | 20 minutes
  Perceived exertion during walking will be quantified every 5 minutes using the OMNI-RES scale.
  Units: Points (0-10).
Adverse effects | 20 minutes
  Severity of adverse sensations (e.g., tingling, burning, numbness, fatigue, discomfort, petechiae) potentially associated with BFR will be recorded.
  Units: Points (0-5).
Affective Responses | 20 minutes
  Affective valence during the exercise bout will be assessed using the Visual Analogue Feeling Scale.
  Units: Points (-5 to +5).

CONTACTS AND LOCATIONS:
Locations (2):
- Faculty of Sport of University of Porto, Porto, Porto District, Portugal
- Faculty of Education of University of La Laguna, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No